CLINICAL TRIAL: NCT01367470
Title: Effects on Cytokines, Immunoglobulins, Antibodies, Sphingomyelinase and PAF Hydrolysis Capacity in the Maternal Milk After Probiotic VSL#3 Administration in the Last Four Weeks of Gestation and First Month of Lactation
Brief Title: Influence of Probiotic VSL#3 Administration on Metabolic and Immunological Profile of the Milk of Breastfeeding Mothers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Prof. Maria Elisabetta Baldassarre, Professor of Pediatrics, Policlinico Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 486Baldassarre
Record Dates: First submitted 2011-04-15; First posted 2011-06-07 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VSL#3 probiotic preparation (Active Comparator): 30 mothers in the last 4 weeks of gestation and in the first month of breastfeeding will be given (after obtaining their informed consent) 1 sachet per day of probiotics (VSL#3) during the last four weeks of pregnancy and the first month of breastfeeding for four weeks under the usual fasting dosage scheme (1 sachet before meal).
  Interventions: Dietary Supplement: VSL#3 probiotic preparation
- Placebo VSL#3 (Placebo Comparator): 30 mothers in the last 4 weeks of gestation and in the first month of breastfeeding will be given (after obtaining their informed consent) a placebo comparable to VSL#3 during the last four weeks of pregnancy and the first month of breastfeeding for four weeks under the usual fasting dosage scheme (1 sachet/day, before meal)
  Interventions: Other: Placebo VSL#3

INTERVENTIONS:
Dietary Supplement: VSL#3 probiotic preparation — VSL#3 is a mixture of 8 different strains of lactic acid bacteria and bifidobacteria at a concentration of 900 billion bacteria per sachet. The suggested dosage is 1 to 2 sachets per day.
  Other Names: VSL#3
  Arms: VSL#3 probiotic preparation
Other: Placebo VSL#3 — Placebo VSL#3 is a base of corn starch containing no active ingredient.
  Other Names: Placebo
  Arms: Placebo VSL#3

SUMMARY:
The newborn immune system is influenced by maternal immunity through both placenta and breastfeeding.

There exists a close interaction between the mother and the baby during gestation and lactation. Maternal milk contains a number of factors that protect the newborn against infections including 1) cytokines and their receptors which are also thought to play a role in the protection against allergies; 2) oligosaccharides with low molecular weight and 3) probiotic bacteria that contribute to the development of the newborn immune system.

Probiotics have a potent immunogenic activity as well as an immunoprotective potential in maternal milk after administration of probiotics during pregnancy and breastfeeding. In addition probiotics are supposed to play a role in the increased production of sphingomyelinase.

DETAILED DESCRIPTION:
Effects on cytokines, on sphingomyelinase and PAF hydrolysis capacity in the maternal milk of term newborns after maternal probiotics administration in the last four weeks of gestation and/or during the first month of lactation.

The newborn immune system is influenced by maternal immunity through both placenta and breastfeeding.

There exists a close interaction between the mother and the baby during gestation and lactation. Maternal milk contains a number of factors that protect the newborn against infections including 1)cytokines and their receptors which are also thought to play a role (albeit still partially controversial) in the protection against allergies; 2) oligosaccharides with low molecular weight and 3) probiotic bacteria that contribute to the development of the newborn immune system.

Probiotics have a potent immunogenic activity as well as an immunoprotective potential in maternal milk after administration of probiotics during pregnancy and breastfeeding. In addition probiotics are supposed to play a role in the increased production of sphingomyelinase, and other enzymes.

Aim of the study

Assessment of the breast milk of women who delivered healthy term babies, as well as of other parameters including the immunomodulatory effect, sphingomyelinase concentration and PAF hydrolysis capacity after administration of the probiotic VSL#3 (VSL Pharmaceuticals) to the mothers in the last four weeks of gestation and in first month of breastfeeding.

Controlled Blind Prospective Study. Group 1 (maternal milk/ cases): 30 mothers in the last four weeks of gestation and in the first month of breastfeeding. All mothers will be given (after obtaining their informed consent) probiotics (VSL#3) during the last four weeks of pregnancy and the first month of breastfeeding under the usual dosage scheme (1 sachet/day, before meal); Group 2 (maternal milk/controls): 30 mothers in the last for weeks of gestation and in the first month of breastfeeding. These mothers will not be given the probiotics in question.

Groups 1 and 2 will undergo assessment of the concentrations of immunoglobulins (secretory IgA), TGF-beta, IL 10 e IL 6, as well as assessment of sphingomyelinase and PAF hydrolysis capacity in colostrum (3-4 days of lactation), in transition milk (1st week of lactation), in mature milk (after the 1st week of lactation) and at the end of the first month of lactation. The samples will be analyzed for the probiotic microorganisms. Furthermore, in parallel, metabolic profiles by 1HNMR spectroscopy will be performed on the same samples of colostrum, transition and mature milk.

The same cytokines, immunoglobulins, sphingomyelinase and PAF hydrolysis capacity and microbiota will be then assessed in the faeces of the newborns on the same days.

The data of each subject enrolled in the study will be collected in Data Sheet which will also include the assessment of the mother's risk of allergy.

A Data Sheet will also be envisaged for each newborn enrolled in the study which will also include daily assessments of gastric stagnation, vomit episodes and abdominal distension.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* able to give informed consent

Exclusion Criteria:

* twin pregnancies, pregnancy diseases (threat of miscarriage, maternal chronic conditions)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2010-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Effect of VSL#3 probiotic administration on breast milk | 2 months
  Assessment of the effects of administration of a probiotic in the last four weeks of gestation and/or during the first month of lactation on the breast milk concentrations of cytokines (TGF-beta, IL-6, IL-10) and immunoglobulines (IGG, IGA, IGM) as well as metabolic profiles and the amount of probiotic species. A total of 30 mothers per arm is expected to be enrolled in the study. Interim analysis will be conducted upon completion of 9 patients per arm.

SECONDARY OUTCOMES:
Assessment of sphingomyelinase concentration in breastmilk of mothers | 2 months
Assessment of PAF hydrolysis in breastmilk of mothers | 2 months
Assessment of fecal newborn microbiota | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Maria Elisabetta Baldassarre, PhD, Principal Investigator — Bari University
Locations (2):
- Italy (2):
  - Dept Of Obstetrics and Neonatology - Section of Neonatology University of Bari Policlinico Hospital, Bari
  - to Be Confirmed, Bari

REFERENCES:
- [Derived] Crepinsek MA, Taylor EA, Michener K, Stewart F. Interventions for preventing mastitis after childbirth. Cochrane Database Syst Rev. 2020 Sep 29;9(9):CD007239. doi: 10.1002/14651858.CD007239.pub4. PMID 32987448
- [Derived] Vitali B, Cruciani F, Baldassarre ME, Capursi T, Spisni E, Valerii MC, Candela M, Turroni S, Brigidi P. Dietary supplementation with probiotics during late pregnancy: outcome on vaginal microbiota and cytokine secretion. BMC Microbiol. 2012 Oct 18;12:236. doi: 10.1186/1471-2180-12-236. PMID 23078375